CLINICAL TRIAL: NCT03071393
Title: Acute Intermittent Hypoxia to Enhance Motor Function After Spinal Cord Injury
Brief Title: Intermittent Hypoxia to Enhance Motor Function After Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201601680
Record Dates: First submitted 2017-02-20; First posted 2017-03-06 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2021-12

CONDITIONS: Spinal Cord Injuries
Keywords: acute intermittent hypoxia; breathing; spinal cord injury; motor function
MeSH Terms: conditions — Spinal Cord Injuries; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects will be asked to participate in two visits at least 7 days apart. Subjects will be assessed on various clinical outcomes before and after an exposure to one of two treatments. In one visit, subjects will be assessed before and after acute intermittent hypoxia, consisting of brief exposures of breathing low oxygen air, alternated with brief exposures to room air. In the other visit, subjects will be assessed before and after an exposure to a sham treatment, consisting of breathing brief exposures of normal oxygen air, alternated with brief exposures to room air. Subjects will undergo acute intermittent hypoxia or a sham treatment in a randomized order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Acute Intermittent Hypoxia, then Sham Intermittent Hypoxia (Experimental): Subjects with chronic spinal cord injury first received an acute intermittent hypoxia protocol with low oxygen air (9-15% inspired oxygen). After a washout period of at least one week, they then received sham intermittent hypoxia with normal oxygen air (21% inspired oxygen).
  Interventions: Device: Hypoxia via Hypoxico Hyp-123; Device: Sham via Hypoxico Hyp-123
- Sham Intermittent Hypoxia, then Acute Intermittent Hypoxia (Experimental): Subjects with chronic spinal cord injury first received a sham (placebo) intermittent hypoxia protocol with normal oxygen air (21% inspired oxygen). After a washout period of at least one week, they then received an acute intermittent hypoxia protocol with low oxygen air (9-15% inspired oxygen).
  Interventions: Device: Hypoxia via Hypoxico Hyp-123; Device: Sham via Hypoxico Hyp-123

INTERVENTIONS:
Device: Hypoxia via Hypoxico Hyp-123 — During acute intermittent hypoxia, subjects will undergo 15 brief exposures (60-120 seconds) of low oxygen air (9-15% inspired oxygen) delivered by an air generator, alternated with 15 brief exposures (60-120 seconds) of ambient room air.
  Other Names: Altitude Generator
Device: Sham via Hypoxico Hyp-123 — During sham intermittent hypoxia, subjects will undergo 15 brief exposures (60-120 seconds) of normal oxygen air (21% inspired oxygen) delivered by an air generator, alternated with 15 brief exposures (60-120 seconds) of ambient room air.
  Other Names: Altitude Generator

SUMMARY:
This study will examine if acute intermittent hypoxia (brief episodes of breathing lower oxygen), which has been shown to enhance plasticity and motor output, can enhance functional outcomes and muscle activation in individuals with spinal cord injury. Our aim is to assess breathing, sitting, standing and walking functional ability before and after acute intermittent hypoxia, compared to a sham treatment. This information may be useful in advancing rehabilitation for people with spinal cord injuries.

DETAILED DESCRIPTION:
Recent evidence has shown that acute intermittent hypoxia can strengthen motor pathways after spinal cord injury, and enhance walking outcomes after walking rehabilitation compared to walking rehabilitation alone. A single session of acute intermittent hypoxia has also been shown to temporarily enhance breathing and limb strength in people with spinal cord injury. Further evidence supports the hypothesis that acute intermittent hypoxia acts on all motor pathways, and thus can enhance the strength of most muscles in the body.

Spinal cord injury affects the muscles that control respiration. Decreased respiratory muscle function can lead to diseases of the respiratory system, which are the primary cause of death and significant cause of re-hospitalization after spinal cord injury. Deficits in postural muscle function affect one's ability to balance, safely maintain a seated position, or ambulate after spinal cord injury, severely impacting daily activities such as self-care and feeding skills.

This study will test the hypothesis that a single session of acute intermittent hypoxia will increase strength and activation of the muscles that control respiration and posture, leading to improved scores on functional assessments in individuals with chronic spinal cord injury. Our long term goal is to better understand the therapeutic potential of acute intermittent hypoxia combined with physical rehabilitation for individuals with chronic spinal cord injury.

ELIGIBILITY:
Inclusion criteria:

1. Male or female, ages 18-65
2. Greater than 6 months post-spinal cord injury
3. Spinal cord injury affecting segments between C4-T12
4. No other known neurological disorders
5. Able to provide informed consent
6. no severe musculoskeletal impairments, open wounds, or skin lesions that would limit participation in functional assessments.

Exclusion criteria:

1. Presence of a self-reported uncontrolled medical condition including, but not limited to: cardiovascular disease; sleep apnea; obstructive lung disease; severe neuropathic or chronic pain; severe recurrent autonomic dysreflexia
2. Severe, untreated bladder or urinary tract infection
3. Presence of severe musculoskeletal impairments, open wounds, or skin lesions that would limit participation in functional assessments
4. Women who report being pregnant or test positive on a pregnancy test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily J Fox, MHS, DPT, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Brooks Rehabilitation, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonzalez-Rothi EJ, Lee KZ, Dale EA, Reier PJ, Mitchell GS, Fuller DD. Intermittent hypoxia and neurorehabilitation. J Appl Physiol (1985). 2015 Dec 15;119(12):1455-65. doi: 10.1152/japplphysiol.00235.2015. Epub 2015 May 21. PMID 25997947
- [Background] Hayes HB, Jayaraman A, Herrmann M, Mitchell GS, Rymer WZ, Trumbower RD. Daily intermittent hypoxia enhances walking after chronic spinal cord injury: a randomized trial. Neurology. 2014 Jan 14;82(2):104-13. doi: 10.1212/01.WNL.0000437416.34298.43. Epub 2013 Nov 27. PMID 24285617
- [Background] Trumbower RD, Jayaraman A, Mitchell GS, Rymer WZ. Exposure to acute intermittent hypoxia augments somatic motor function in humans with incomplete spinal cord injury. Neurorehabil Neural Repair. 2012 Feb;26(2):163-72. doi: 10.1177/1545968311412055. Epub 2011 Aug 5. PMID 21821826
- [Background] Tester NJ, Fuller DD, Fromm JS, Spiess MR, Behrman AL, Mateika JH. Long-term facilitation of ventilation in humans with chronic spinal cord injury. Am J Respir Crit Care Med. 2014 Jan 1;189(1):57-65. doi: 10.1164/rccm.201305-0848OC. PMID 24224903
- [Background] Satriotomo I, Nichols NL, Dale EA, Emery AT, Dahlberg JM, Mitchell GS. Repetitive acute intermittent hypoxia increases growth/neurotrophic factor expression in non-respiratory motor neurons. Neuroscience. 2016 May 13;322:479-88. doi: 10.1016/j.neuroscience.2016.02.060. Epub 2016 Mar 2. PMID 26944605
- [Result] Sutor T, Cavka K, Vose AK, Welch JF, Davenport P, Fuller DD, Mitchell GS, Fox EJ. Single-session effects of acute intermittent hypoxia on breathing function after human spinal cord injury. Exp Neurol. 2021 Aug;342:113735. doi: 10.1016/j.expneurol.2021.113735. Epub 2021 May 2. PMID 33951477

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals were recruited through advertisements and rehabilitation health facilities in north Florida. Recruitment occurred from 07/2017 through 12/2019.
Groups:
- Acute Intermittent Hypoxia, Then Sham Intermittent Hypoxia: Subjects with chronic spinal cord injury first received an acute intermittent hypoxia protocol with low oxygen air (9-15% inspired oxygen). After a washout period of at least one week, they then received sham intermittent hypoxia with normal oxygen air (21% inspired oxygen).
  Hypoxico Hyp-123: During acute intermittent hypoxia, subjects will undergo 15 brief exposures (60-120 seconds) of low oxygen air (9-15% inspired oxygen) delivered by an air generator, alternated with 15 brief exposures (60-120 seconds) of ambient room air.
- Sham Intermittent Hypoxia, Then Acute Intermittent Hypoxia: Subjects with chronic spinal cord injury first received a sham (placebo) intermittent hypoxia protocol with normal oxygen air (21% inspired oxygen). After a washout period of at least one week, they then received an acute intermittent hypoxia protocol with low oxygen air (9-15% inspired oxygen).
  Hypoxico Hyp-123: During sham intermittent hypoxia, subjects will undergo 15 brief exposures (60-120 seconds) of normal oxygen air (21% inspired oxygen) delivered by an air generator, alternated with 15 brief exposures (60-120 seconds) of ambient room air.
Period: First Intervention (Single Day Session)
Arm/Group | Acute Intermittent Hypoxia, Then Sham Intermittent Hypoxia | Sham Intermittent Hypoxia, Then Acute Intermittent Hypoxia
Started | 7 | 10
Completed | 7 | 10
Not Completed | 0 | 0
Period: Washout (at Least 7 Days)
Arm/Group | Acute Intermittent Hypoxia, Then Sham Intermittent Hypoxia | Sham Intermittent Hypoxia, Then Acute Intermittent Hypoxia
Started | 7 | 10
Completed | 7 | 10
Not Completed | 0 | 0
Period: Intervention 2 (Single Day Session)
Arm/Group | Acute Intermittent Hypoxia, Then Sham Intermittent Hypoxia | Sham Intermittent Hypoxia, Then Acute Intermittent Hypoxia
Started | 7 | 10
Completed | 7 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Subjects with chronic spinal cord injury completed a single session of acute intermittent hypoxia with low oxygen air (15 exposures of 60-120 seconds, 9-15% inspired oxygen, alternated with 60-120 seconds of room air) and a single session of sham acute intermittent hypoxia with room air (15 exposures of room air, 60-120 seconds, 21% oxygen). A washout of at least 7 days separated the two sessions.
Arm/Group | All Study Participants
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17
ASIA Impairment Scale [Count of Participants; unit: Participants] — American Spinal Injury Association Impairment Scale to grade injury severity. AIS "A" implies no motor or sensory function below the injury level, and is considered the most severe injury category. AIS "B" implies no motor function but at least partially preserved sensory function below the injury level. AIS "C" implies minimal-to-moderate motor function and at least partially preserved sensory function below the injury. AIS "D" implies minimal deficits in sensory and motor function below the injury, and is considered the least severe injury category.
  Participants
    AIS A Complete SCI | 6
    AIS B motor complete SCI | 7
    AIS C motor incomplete | 3
    AIS D motor incomplete | 1
Spinal Cord Injury chronicity [Mean (Standard Deviation); unit: months] — Time since injury onset in months
  months | 63.1 (112.9)
Upper Extremity Motor Score (UEMS) [Mean (Standard Deviation); unit: units on a scale] — UEMS measures total strength in 5 key upper extremity muscles on both sides. Scores can range from 0 (no preserved strength in upper extremities) to 50 (fully preserved strength in upper extremities).
  units on a scale | 40.2 (15.3)
Lower Extremity Motor Score (LEMS) [Mean (Standard Deviation); unit: units on a scale] — LEMS measures total strength in 5 key lower extremity muscles on both sides. Scores can range from 0 (no preserved strength in lower extremities) to 50 (fully preserved strength in lower extremities).
  units on a scale | 4.6 (12.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximal Inspiratory Pressure
Description: An assessment of inspiratory muscle strength.
Time Frame: Change between baseline and 30 minutes post-intermittent hypoxia or sham.
Population: All participants completed the measure and were analyzed
Measure: Mean (Standard Deviation); unit: cmH2O
Groups:
- All Study Participants - Acute Intermittent Hypoxia: Subjects with chronic spinal cord injury completed a single session of acute intermittent hypoxia with low oxygen air (15 exposures of 60-120 seconds, 9-15% inspired oxygen, alternated with 60-120 seconds of room air) Individuals were 13 males; 34.1 ± 14.5 years old; 13 motor complete SCI; >6 months post injury
- All Study Participants - Sham: Subjects with chronic spinal cord injury completed a single session of acute sham intermittent hypoxia with room air Individuals were 13 males; 34.1 ± 14.5 years old; 13 motor complete SCI; >6 months post injury
Arm/Group | All Study Participants - Acute Intermittent Hypoxia | All Study Participants - Sham
Number analyzed (Participants) | 17 | 17
cmH2O | 8.2 (12.3) | -3.0 (11.3)
Statistical Analysis 1: Comparison: All Study Participants - Acute Intermittent Hypoxia vs All Study Participants - Sham; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Maximal Expiratory Pressure
Description: An assessment of expiratory muscle strength.
Time Frame: Change between baseline and 30 minutes post-intermittent hypoxia or sham.
Population: All participants completed the measure and were analyzed
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | All Study Participants - Acute Intermittent Hypoxia | All Study Participants - Sham
Number analyzed (Participants) | 17 | 17
cmH2O | 4.3 (11.5) | 2.9 (9.8)
Statistical Analysis 1: Comparison: All Study Participants - Acute Intermittent Hypoxia vs All Study Participants - Sham; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Change in Forced Vital Capacity
Description: An assessment of how much air a person can forcefully exhale after a maximal inspiratory effort.
Time Frame: Change between baseline and 30 minutes post-intermittent hypoxia or sham.
Population: The measure was not obtained on 3 participants
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- All Study Participants - Acute Intermittent Hypoxia: Subjects with chronic spinal cord injury completed a single session of acute intermittent hypoxia with low oxygen air (15 exposures of 60-120 seconds, 9-15% inspired oxygen, alternated with 60-120 seconds of room air)
- All Study Participants - Sham: Subjects with chronic spinal cord injury completed a single session of acute sham intermittent hypoxia with room air
Arm/Group | All Study Participants - Acute Intermittent Hypoxia | All Study Participants - Sham
Number analyzed (Participants) | 14 | 14
Liters | -0.01 (0.17) | 0.00 (0.21)
Statistical Analysis 1: Comparison: All Study Participants - Acute Intermittent Hypoxia vs All Study Participants - Sham; Test type: Superiority; p < 0.05, ANOVA

4. Primary Outcome: Change in Mouth Occlusion Pressure (P0.1)
Description: An assessment of the pressure generated in the first 0.1 seconds of the participant's initiation of inhalation.
Time Frame: Change between baseline and 30 minutes post-intermittent hypoxia or sham.
Population: This measure was obtained in 12 participants. 12 participants were analyzed.
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | All Study Participants - Acute Intermittent Hypoxia | All Study Participants - Sham
Number analyzed (Participants) | 12 | 12
cmH2O | 0.24 (0.30) | 0.15 (0.50)
Statistical Analysis 1: Comparison: All Study Participants - Acute Intermittent Hypoxia vs All Study Participants - Sham; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney) — Uncorrected p values are reported

ADVERSE EVENTS:
Time Frame: 3 weeks
Description: The study was low risk and there were no adverse events. Participants were monitored for safety as described in the protocol. As required, a cumulative adverse event table was submitted annually to the IRB.
Groups:
- Acute Intermittent Hypoxia: Subjects with chronic spinal cord injury will undergo an acute intermittent hypoxia protocol with low oxygen air (9-15% inspired oxygen.
  Hypoxico Hyp-123: During acute intermittent hypoxia, subjects will undergo 15 brief exposures (60-120 seconds) of low oxygen air (9-15% inspired oxygen) delivered by an air generator, alternated with 15 brief exposures (60-120 seconds) of ambient room air.
- Sham Intermittent Hypoxia: Subjects with chronic spinal cord injury will undergo a sham placebo protocol with normal oxygen air (21% inspired oxygen).
  Hypoxico Hyp-123: During sham intermittent hypoxia, subjects will undergo 15 brief exposures (60-120 seconds) of normal oxygen air (21% inspired oxygen) delivered by an air generator, alternated with 15 brief exposures (60-120 seconds) of ambient room air.
Arm/Group | Acute Intermittent Hypoxia | Sham Intermittent Hypoxia
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/93/NCT03071393/Prot_SAP_000.pdf